CLINICAL TRIAL: NCT04322123
Title: An Open-label, Randomized Controlled Trial of Hydroxychloroquine and Azithromycin for COVID-19 Infection on Hospitalized, Noncritical Patients
Brief Title: Safety and Efficacy of Hydroxychloroquine Associated With Azithromycin in SARS-Cov-2 Virus (COVID-19)
Acronym: Coalition-I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: Hospital Israelita Albert Einstein (Other); Hospital Sirio-Libanes (Other); Brazilian Research In Intensive Care Network (Network); EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Brazil COVID Coalition I Trial
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Coronavirus Infections
MeSH Terms: conditions — Coronavirus Infections | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydroxychloroquine (Experimental): Hydroxychloroquine after randomization, Hydroxychloroquine [400mg 2x/day, 12/12h] for 07 days.
  Interventions: Drug: Hydroxychloroquine Oral Product
- Hydroxychloroquine + azithromycin (Experimental): Hydroxychloroquine + azithromycin. After randomization, Hydroxychloroquine [400mg 2x/day, 12/12h] + azithromycin [500mg 1x/day]) for 07 days.
  Interventions: Drug: Hydroxychloroquine + azithromycin
- Control (No Intervention): standard treatment protocol for 2019-nCoV infection.

INTERVENTIONS:
Drug: Hydroxychloroquine Oral Product — Hydroxychloroquine 400 mg BID
  Arms: Hydroxychloroquine
Drug: Hydroxychloroquine + azithromycin — Hydroxychloroquine 400 mg BID + azithromycin 500 mg once a day
  Arms: Hydroxychloroquine + azithromycin

SUMMARY:
Coronavirus (COVID-19) is a somewhat new and recognized infectious disease that is now spreading to several countries in the world, including Brazil. Hydroxychloroquine and azithromycin may be useful for treating those patients.

COALITION I study aims to compared standard of care, hydroxychloroquine plus azithromycin and hydroxychloroquine monotherapy for treatment of hospitalized patients with COVID-19.

COALITION I will recruit 630 patients with infection by COVID-19 (210 per arm). Ordinal endpoint of status at 15 days will be the primary endpoint.

DETAILED DESCRIPTION:
The current pandemic associated with coronavirus disease 2019 (COVID-19) represents a major global health challenge. There are no effective therapies for the management of COVID-19 that have been proven to improve clinical outcomes in this high-risk group of patients. Hydroxychloroquine and its combination with azithromycin have been suggested to improve viral clearance, but its effect on clinical outcomes remains uncertain.

This is an open-label pragmatic multicentre randomized (concealed) clinical trial of 7 days of hydroxychloroquine (400 mg BID) plus azithromycin (500 mg once daily), hydroxychloroquine 400 mg BID, or standard of care for moderately severe hospitalized patients with suspected or confirmed COVID-19 (in-patients with up to 4L/minute oxygen supply through nasal catheter). Patients are randomized in around 50 recruiting sites (630 patients with confirmed COVID-19; 1:1:1; 210 patients per arm).

The primary endpoint is a 7-level ordinal scale measured at 15-days: 1) not hospitalized, without limitations on activities; 2) not hospitalized, with limitations on activities; 3) hospitalized, not using supplementary oxygen; 4) hospitalized, using supplementary oxygen; 5) hospitalized, using high-flow nasal cannula or non-invasive ventilation; 6) hospitalized, on mechanical ventilation; 7) death. Secondary endpoints are the ordinal scale at 7 days, need for mechanical ventilation and rescue therapies during 15 days, need of high-flow nasal cannula or non-invasive ventilation during 15 days, length of hospital stay, in-hospital mortality, thromboembolic events, occurrence of acute kidney injury, defined as an increase in creatinine above 1.5 times the baseline value and number of days free of respiratory support at 15 days. Secondary safety outcomes include prolongation of QT interval on electrocardiogram, ventricular arrhythmias, and liver toxicity. The main analysis will consider all patients with confirmed COVID-19 in the groups they were randomly assigned.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected or confirmed COVID-19 admitted to inpatient units and intensive care units

Exclusion Criteria:

* Need for oxygen supplementation > 4 litters per min
* Patients using a high-flow nasal catheter
* Patients using non-invasive mechanical ventilation
* Patients using invasive mechanical ventilation
* Males and females aged < 18 years
* Pregnancy
* Allergy to chloroquine or derivatives
* Allergy to azithromycin
* Patients that have already received more than one dose of either azithromycin or hydroxychloroquine before enrollment
* Patients with respiratory symptoms for more than 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of the clinical status | 15 days after randomization
  Evaluation of the clinical status of patients on the 15th day after randomization defined by the Ordinal Scale of 7 points.
  1. Alive at home without limitations on activities
  2. Alive at home without limitations on activities
  3. In the hospital without oxygen
  4. In the hospital using oxygen
  5. In the hospital using high-flow nasal catheter or non-invasive ventilation
  6. In hospital, on mechanical ventilation
  7. Dead

SECONDARY OUTCOMES:
Ordinal scale in 7 days | 7 days after randomization
  Evaluation of the clinical status of patients on the 7th day after randomization defined by the Ordinal Scale of 7 points.
  1. Alive at home without limitations on activities
  2. Alive at home without limitations on activities
  3. In the hospital without oxygen
  4. In the hospital using oxygen
  5. In the hospital using high-flow nasal catheter or non-invasive ventilation
  6. In hospital, on mechanical ventilation
  7. Dead
Need of intubation and mechanical ventilation | 7 days after randomization
  Need of intubation and mechanical ventilation up to the 7th day after randomization
Use of mechanical ventilation during hospital stay | 15 days after randomization
  Use of mechanical ventilation during hospital stay
Use of non-invasive ventilation | 7 days after randomization
  Use of non-invasive ventilation up to the 7th day after randomization
Hospital Length of Stay | 28 days after randomization
  Hospital Length of Stay
All-cause mortality | 28 days after randomization
  All-cause mortality rates during hospital stay
Thromboembolic complications | 15 days after randomization
  Occurrence of thromboembolic complications such as:
  Deep vein thrombosis Pulmonary Embolism Stroke
Acute renal disfunction | 15 days after randomization
  Occurrence of renal dysfunction, defined as an increase in creatinine above 1.5 times the baseline value
Number of days alive and free of respiratory support up to 15 days | 15 days
  Number of days alive and free of respiratory support up to 15 days (DAFOR15), defined as the sum of days patients did not require supplementary oxygen, non-invasive ventilation, high-flow nasal catheter neither mechanical ventilation at 15 -days. Patients that perished during the 15-day window will receive zero DAFOR15.

OTHER OUTCOMES:
Safety outcome on corrected QT interval | At day 3 and 7 after enrollment
  Corrected QT interval

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Biasi, PhD, Study Chair — Hospital do Coração; Otavio Berwanger, Principal Investigator — Hospital Israelita Albert Einstein
Locations (28):
- Brazil (28):
  - Hospital Maternidade São José - UNESC - Fundação Social Rural de Colatina, Colatina, Espírito Santo
  - Hospital Geral Clériston Andrade, Feira de Santana, Estado de Bahia
  - Hospital Ana Nery - HAN/SESAB, Salvador, Estado de Bahia
  - HHospital SAMUR, Vitória da Conquista, Estado de Bahia
  - Hospital Geral de Vitória da Conquista, Vitória da Conquista, Estado de Bahia
  - Hospital de Brasília, Brasília, Federal District
  - Instituto de Cardiologia do Distrito Federal, Brasília, Federal District
  - Hospital Vila da Serra, Nova Lima, Minas Gerais
  - Santa Casa de Misericórdia de São João Del Rei, São João del Rei, Minas Gerais
  - Associação Evangélica Beneficente de Londrina - Hospital Evangélico de Londrina, Londrina, Paraná
  - Instituto Estadual do Cérebro Paulo Niemeyer, Rio de Janeiro, Rio de Janeiro
  - Hospital Geral de Caxias do Sul, Caxias do Sul, Rio Grande do Sul
  - Hospital Santa Rita - Irmandade Santa Casa de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Francisco - Irmandade Santa Casa de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São José, Criciúma, Santa Catarina
  - Hospital Baía Sul - Baía Sul Medical Center, Florianópolis, Santa Catarina
  - Hospital Nereu Ramos, Florianópolis, Santa Catarina
  - Centro Hospitalar Unimed, Joinville, Santa Catarina
  - Hospital SEPACO, São Paulo, S
  - Hospital de Amor - Unidade Barretos (Fundação PIO XII), Barretos, São Paulo
  - Casa de Saúde Santa Marcelina, São Paulo, São Paulo
  - Hospital Albert Einstein, São Paulo, São Paulo
  - Hospital Beneficência Portuguesa - Real e Benemérita Associação Portuguesa de Beneficência, São Paulo, São Paulo
  - Hospital BP Mirante - Real e Benemérita, São Paulo, São Paulo
  - Hospital das Clínicas da FMUSP, São Paulo, São Paulo
  - Hospital do Servidor Público Estadual - HSPE - IAMSPE, São Paulo, São Paulo
  - Hospital São Paulo - UNIFESP, São Paulo, São Paulo
  - Hospital Sírio-Libanês, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Furtado RHM, Barros E Silva PGM, Fonseca HAR, Serpa-Neto A, Correa TD, Guimaraes HP, Pereira AJ, Olivato GB, Zampieri FG, Lisboa T, Junqueira DLM, Lapa MG, Monfardini F, Damiani LP, Echenique LS, Gebara OE, Hoffman Filho CR, Polanczyk CA, Rohde LE, Amazonas R, Machado FR, Avezum A, Azevedo LCP, Veiga VC, Rosa RG, Lopes RD, Cavalcanti AB, Berwanger O; COALITION COVID-19 Brazil Steering Committee and Investigators. Cardiovascular Safety of Azithromycin in Patients Hospitalized With COVID-19: A Prespecified Pooled Analysis of the COALITION I and COALITION II Randomized Clinical Trials. Am J Cardiol. 2024 Mar 1;214:18-24. doi: 10.1016/j.amjcard.2023.11.069. Epub 2023 Dec 15. PMID 38104755
- [Derived] Cavalcanti AB, Zampieri FG, Rosa RG, Azevedo LCP, Veiga VC, Avezum A, Damiani LP, Marcadenti A, Kawano-Dourado L, Lisboa T, Junqueira DLM, de Barros E Silva PGM, Tramujas L, Abreu-Silva EO, Laranjeira LN, Soares AT, Echenique LS, Pereira AJ, Freitas FGR, Gebara OCE, Dantas VCS, Furtado RHM, Milan EP, Golin NA, Cardoso FF, Maia IS, Hoffmann Filho CR, Kormann APM, Amazonas RB, Bocchi de Oliveira MF, Serpa-Neto A, Falavigna M, Lopes RD, Machado FR, Berwanger O; Coalition Covid-19 Brazil I Investigators. Hydroxychloroquine with or without Azithromycin in Mild-to-Moderate Covid-19. N Engl J Med. 2020 Nov 19;383(21):2041-2052. doi: 10.1056/NEJMoa2019014. Epub 2020 Jul 23. PMID 32706953
- Available data/document: Study Protocol — https://www.medrxiv.org/content/10.1101/2020.05.19.20106997v1 — Preprint of the Protocol